CLINICAL TRIAL: NCT03922867
Title: Comparison of Feasibility and Efficacy of a Web-based Cognitive Behavioral Therapy Versus Usual Care for Management of Insomnia in Patients With Fibromyalgia
Brief Title: Web-based CBT for Insomnia Patients With Fibromyalgia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Ravindra Ganesh, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 18-011637
Record Dates: First submitted 2019-04-18; First posted 2019-04-22 (Actual); Last update posted 2021-03-05 (Actual); Status verified 2021-03

CONDITIONS: Insomnia; Fibromyalgia
Keywords: insomnia; fibromyalgia
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Fibromyalgia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention): Subjects with receive standard of care for management of insomnia in subjects with fibromyalgia
- Intervention Group (Active Comparator): Subjects will receive standard of care and additionally complete the online cognitive behavior therapy program
  Interventions: Behavioral: CBT

INTERVENTIONS:
Behavioral: CBT — A web-based educational platform to deliver cognitive behavioral therapy (CBT) for insomnia
  Arms: Intervention Group

SUMMARY:
Researchers are evaluating if cognitive behavioral therapy for insomnia delivered over the internet will help with fibromyalgia symptoms.

DETAILED DESCRIPTION:
The investigators are studying the effect of an internet-based cognitive behavioral therapy for insomnia, compared with usual care in fibromyalgia patients. Fibromyalgia patients will consent to study, and a determination made if the patients meet criteria. If eligible, qualifying patients will be randomized, and begin participation in randomized intervention. During participation on the study subjects will complete surveys at set intervals.

ELIGIBILITY:
Inclusion Criteria:

* Meets diagnostic criteria for fibromyalgia
* Has insomnia
* Have internet access and a device that can access the web-based program.

Exclusion Criteria:

* Active sleep disorder which is not treated (obstructive sleep apnea, obesity hypoventilation syndrome)
* Active psychiatric disorder (Bipolar affective disorder, anxiety, depression, schizophrenia) which is not optimally managed.
* Chronic fatigue syndrome
* Morbid obesity

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2019-12-03 (Actual); Primary Completion 2021-02-28 (Actual); Study Completion 2021-03-03 (Actual)

PRIMARY OUTCOMES:
Change in insomnia severity | through study completion, an average of 12 weeks
  Surveying the changes in insomnia severity seen during the subjects participation in the study
Change in attitude towards sleep | through study completion, an average of 12 weeks
  Surveying the subjects attitude towards sleep over the duration of their participation in the study.

SECONDARY OUTCOMES:
Change in fibromyalgia symptoms | through study completion, an average of 12 weeks
  Surveying the change in fibromyalgia symptoms that occur during study participation

CONTACTS AND LOCATIONS:
Overall Officials: Ravindra Ganesh, MBBS, MD, Principal Investigator — Mayo Clinic; Sanjeev Nanda, MD, Study Chair — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials